CLINICAL TRIAL: NCT04701294
Title: Evaluation of the Retention of a Sealant Based on Flowable Resin With Sprg and Another Based on Flowable Resin in First Permanent Molars:Randomized Controlled Clinical Trial in 12 Months
Brief Title: Retention of Flowable Resin With Sprg and of a Flowable Resin in First Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catherine Christie Ruiz Yasuda (Other)
Responsible Party: Sponsor-Investigator, Catherine Christie Ruiz Yasuda, Doctor Catherine Christie Ruiz Yasuda, National University of San Marcos, Peru
Organization: National University of San Marcos, Peru (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0647-FO-UPG-20
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pit and Fissure Sealant
Keywords: pit and fissure sealant; glass ionomer; resin
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Intervention Model Description: A split mouth (120 teeth) study design will be adopted (19.20), which consists of a simple division of the mouth into two parts (right and left) for the first four permanent molars of each patient, where the placement of the materials will be on the right / left side of the mouth and contralateral.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Regarding the patient data, it will only be handled by the programmer who will be in charge of coding, randomizing the first permanent molars, randomizing the materials to be used so that it is placed in the first permanent molars and this information will be given to the coordinator so that the put in sealed envelopes and then these sealed envelopes will be given to an outside assistant so that such data is not disclosed or published.
  Assistant 3 (in charge of labeling with kraft paper and listing the intervention material(giomer F03 beautifil-shofu and Tetric N-Flow ivoclar vivadent) with the research coordinator.
  The evaluators did not do the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giomer Beautifil flow plusF03 Shofu-Japan (Experimental): Giomer beautifil flow plusF03 shofu-Japan an application of flowable resin with sprg as a sealant for pits and fissures on the occlusal surface of permanent first molars until the end of the experiment.
  Interventions: Device: Giomer Beautifil flow plusF03 Shofu-Japan
- Tetric N flow ivoclar vivadent-Germany (Active Comparator): Tetric N flow ivoclar vivadent-Germany an application of flowable resin a sealant for pits and fissures on the occlusal surface of permanent first molars until the end of the comparator.
  Interventions: Device: Tetric N flow ivoclar vivadent-Germany

INTERVENTIONS:
Device: Giomer Beautifil flow plusF03 Shofu-Japan — A pair of permanent first molars will be used for each participant homologs The operator will apply in the upper / lower first molars the sealant material in the order assigned according to the previous randomization. For the intervention group, they will be sealed based on a fluid resin with s-prg glass ionomer filling (Giomer F03 Beautiful -Shofu) in association with a bottle of adhesive (Single Bond) . The evaluation and monitoring process; another operator will record the retention of the sealant in a period of 6, 9 and 12 months.
  Other Names: Experimental
  Arms: Giomer Beautifil flow plusF03 Shofu-Japan
Device: Tetric N flow ivoclar vivadent-Germany — And on the contralateral side (control) the first upper / lower molars will be sealed will be sealed with a fluid resin compound (Tetric N-Flow ivoclar vivadent) in association with a bottle of adhesive (Single Bond). Both materials have a similar color. The operator and the child will not be informed about the brand of the material used. The assistant will collect the data in the file. The evaluation and monitoring process; another operator will record the retention of the sealant in a period of 6, 9 and 12 months.
  Other Names: Control
  Arms: Tetric N flow ivoclar vivadent-Germany

SUMMARY:
Objective: Determine which of the two sealants has better retention during the periods of 6, 9 and 12 months, one based on flowable resin with sprg or the other only based on flowable resin and we have the following hypothesis: the retention of the sealant based on a flowable resin with sprg is greater than a sealant based on a flowable resin in permanent first molars at different periods ".

Materials and methods: 60 children from the school in the district of Pichanaki, Peru and aged 6 to 8 years were included in this study. The Split mouth design will be adopted, and 120 permanent first molars are designated.It will be applied on the upper / lower first molars with sealant material being the order assigned according to the previous randomization, for the intervention group they will be sealed based on flowable resin with sprg (giomer F03 beautifil-Shofu) in association with a bottle of adhesive (single bond) and on the contralateral side the upper / lower first molars will be sealed, the control group will be sealed with a flowable resin-based resin compound (Tetric N-Flow ivoclar vivadent) in association with a bottle of adhesive (Single Bond). Placement of materials on the right / left side of the mouth will be randomly assigned following block randomization procedures with a 1:1 allocation using the random block sizes of 4 and 8 (35).A computerized random number generator will be used. A total of 120 upper / lower molar teeth will be sealed with both materials (60 teeth for each material). The materials will be placed by the same operator according to the protocol of UNMSM for the sealing of pits and deep fissures; then, the interventional group will be compared after a 12-month follow-up with controls at 6, 9 and 12 months. The statistical analysis will be with SPSS software 20.0. Since all the data in this study will be categorical, nonparametric statistics will be used. Expected result: After the evaluation period it is expected to find significant differences in the retention of the sealant to flowable resin base with sprg (giomer F03 beautifil -Shofu) and sealant based on flowable resin (Tetric N- Flow ivoclar vivadent) using an adhesive system . Conclusion: Identify and quantify the retention of a sealant based on flowable resin with sprg (giomer F03 Beautifil -Shofu) and a sealant based on flowable resin (Tetric N-Flow ivoclar vivadent) using an adhesive system on 12 months.

DETAILED DESCRIPTION:
The following research project is being carried out following the 2010 Consort Declaration (32)

1. Ethical considerations: Declaration of Helsinki. Access to the data of the research subjects in order to guarantee their confidentiality according to national regulations and international recommendations .
2. Sample selection In case of natural phenomena, health emergency and the population cannot continue, another population will have to be found. Biosecurity in Sarv-cov2.Recommendations for the Treatment of Pit and Fissure Sealants (36-38)
3. Data collection techniques: Phase 1. Coordination with the Ethics and Parental Authorization Committee The Research Ethics Committee of the Institute of Tropical Medicine Daniel Alcides Carrión UNMSM will give us the first pass. Letters of invitation will be made and they will be distributed in class through the teachers, and each student will take it home to deliver to their parents or guardians; Each letter (envelope) will have the informed consent (Annex 1), the informed consent (Annex 2), data record sheet (Annex 3) and an informative bulletin (Annex 4) where it explains all the procedure that will be carried out for each participant, there will also be an informative talk at the school for parents and teachers, where they will be informed about the study and will collect the envelopes. Research will not force any child to participate; each will have the option of choosing to participate in the study by verbal assent. A report will be delivered to the parent or guardian of the child after the intervention. Informed consent process Researcher 1 will give an informative talk about the study and will collect the envelopes containing the informed consent, informed consent and data record sheet). Students and parents who accept participation will receive a summons for subsequent dental visits (Annex 5). It will collect the consents signed by both parents / guardians and in the event that the signature of one of the parents cannot be obtained either due to impossibility (death, difficulty in obtaining the signature, absence and reasons of personal strength)(39)Only the signature of one will be accepted to give consent; and informed assent if the child reports that he understands and is mature enough to understand(39). Diagnostic Process Assistant 1 will be in charge of bringing the students for their dental check-up and will also provide the materials to operator 1 who will do the oral hygiene and prophylaxis index procedure. Afterwards, operator 2, who has 10 years of experience, will be previously calibrated according to the ICDAS II criteria, using the visual method, he will detect and classify the lesions according to the International System criteria. Detection and Evaluation of Caries (ICDAS-II) (26) and the teeth that will represent scores 0 and 1 will be selected. The inclusion and exclusion criteria mentioned above will be taken into account; and patients who have at least one pair of homologous permanent first molars that meet the same requirements will be considered. The assistant 2 will be in charge of filling in the data sheets of the participants. Operator 1 will evaluate the Simplified Oral Hygiene Index until you reach an OHS score of 1 over a period of one month. Researcher 1 will select the participants taking into account the inclusion and exclusion criteria and will deliver the list of those participants to the programmer for randomization. Treatment randomization process The name of each participant will be coded by letters, this will be done by the programmer; the materials are going to be coded by number and the cards are going to be worked with these codings for their subsequent data analysis. And regarding patient data, it will only be handled by the programmer who will be in charge of coding, randomizing the first permanent molars, randomizing the materials to be used so that it is placed in the first permanent molars and this information will be given to the coordinator so that the put in sealed envelopes and then these sealed envelopes will be given to a housekeeper so that said data is not disclosed or published. In case this section of data confidentiality is in the informed consent it could be mentioned. The programmer will give the randomized list to the coordinator and the coordinator will give the external assistant who is not participating in the clinical trial in sealed envelopes labeled by each participant. This external assistant will bring the randomized patient for treatment. Allocation concealment mechanism process and implementation The programmer without participation in the clinical trial will do the randomization sequence generating the list of numbers randomly assigned to participants and will be created with Stata 16 statistical software (Stata Corp. College Station, TX). The investigators will give this list to the coordinator and this external assistant will receive the envelopes and will take care of taking the patient to receive treatment. Blinding process Blinding will be strictly maintained; by emphasizing it on the operators, assistants, evaluators, workers of the educational institution and the parents / guardians and participants. While the participants, operators, evaluators, assistants assigned to carry out the diagnosis, procedure and placement of the material, will not know the brand of the pit and fissure sealant, due to which will be covered with kraft paper, labeled and numbered .Outcome assessors and data analysts will be blinded to allocation. "The investigators who performed the intervention procedure will not take any result measures. Procedures process Assistant 3 will be in charge of labeling with kraft paper and listing the intervention material A and B (giomer F03 beautifil-Shofu and Tetric N-Flow ivoclar vivadent) in prior coordination with the research coordinator. Operator 3 and assistant 4 will be previously trained and calibrated; they will do the procedure, without knowing the names of the sealants.A split-mouth study design will be used and will be used as follows; It will be applied on the upper / lower first molars with sealing material, being the order assigned according to the previous randomization, for the intervention group they will be sealed based on fluid resin s-prg (giomer F03 beautifil-Shofu) in association with a bottle of adhesive (single bond) and on the contralateral side, the upper / lower first molars will be sealed, the control group will be sealed with a fluid resin compound based on flowable resin (TetricN-Flow ivoclar vivadent) in association with a bottle of adhesive (Single Bond). Placement of materials on the right / left side of the mouth will be randomly assigned following block randomization procedures with a 1:1 allocation using the random block sizes of 4 and 8(35). A computerized random number generator will be used. A total of 120 upper / lower molar teeth will be sealed with both materials (60 teeth for each material). The materials will be placed by the same operator according to the protocol UNMSM for the sealing of pits and deep fissures. Steps for the application of the sealant, the teeth will be isolated with cotton rolls carefully and the assistants 4 will hold a plastic saliva ejector to avoid contamination of the saliva and facilitate the operative procedures of the occlusal surfaces of the upper molars and / or lower for each operator: The occlusal surfaces will be cleaned using water, brush and low hand piece; wash and dry of the occlusal surface; then deproteinization will be done with sodium hypochlorite (5.25%) for 60 seconds, wash with a water / air spray for 30 seconds; and dry. The tooth will then be etched using a 37% orthophosphoric acid gel for 15 seconds, rinsed with a water / air spray for 30 seconds, and dried with cotton balls. For the intervention, the sealants will be covered and listed on Kraft paper, it will be sealed for the intervention fluid resin with sprg (giomer F03 beautifil-Shofu) and for the control group it will be sealed with fluid resin (Tetric N- Flow). Subsequently, a uniform layer of fluid composite resin will be applied and it will be light-cured for 11 seconds using an LED curing unit with an output of 1500 mW / cm2 (Gnatus). The cotton rolls and plastic saliva ejector will be removed, and the occlusion will be checked with articulating paper. The operator will not know the brand of sealant to be used, because it will be covered with Kraft paper and will be delivered by another person(assistant) previously trained for this activity and both materials have a similar color. The child will also not be informed about the brand of the material used. The assistant 5 will collect the data on the card. An average attendance will be 6 participants per day with time intervals to prepare the work environment between each procedure. Evaluation and monitoring process: Assistant 6 will bring and take the participants to operator 4 who will do the prophylaxis and help fill out the cards. Operator 5 with at least ten years of experience it will be previously trained, evaluated and calibrated; in accordance with ICDAS-S II criteria and retention of sealants. The calibration will be given by the Kappa measure (κ >0.7). Operator 5 will not have performed the pit and fissure sealants procedure, he will record the retention of the sealant in a period of 6, 9 and 12 months. Follow-up of sealed teeth will be observed in good lighting, after tooth prophylaxis. Evaluation will be performed with an oral mirror and periodontal probe. Each sealant is classified as follows: Total retention of the sealant in all pits and fissures (RT). Partial retention of sealant in some pits and fissures (PP). Total loss of sealant in all pits and fissures (TP): no trace of materials is detected on the surface. The coordinator will be in all the evaluation follow-ups. Statistical process The Statesman informs the coordinator of the tooth coding and materials. Phase 2. Calibration The researcher who will diagnose and apply the pit and fissure sealants will be trained by a principal teacher the Universidad Nacional Mayor de San Marcos, calibrated in ICDAS II and in Minimal Intervention Dentistry. Phase 3. Pilot Study The pilot phase had the purpose of planning and organizing the study, measuring work time, the four-hand technique, preparing the materials for treatment (covering the sealants with a Kraft paper), recording the information and the evaluation in controls. This pilot will take place in the Juan Pablo Vizcardo y Guzmán School.

ADVERSE EVENTS A. THE PROCEDURES FOR OBTAINING, RECORDING AND MONITORING ADVERSE EVENTS BY THE INVESTIGATOR AND THEIR NOTIFICATION TO THE SPONSOR The investigators have a registration form that is in annex 11 and that will be monitored at 6, 9 and 12 months, the investigators will be in constant communication with the school and parents and / or guardians will be able to communicate and this information is in the Appendix 1.It is important to remember that the rights, welfare and safety of research participants will always prevail over the interests of science and society. Therefore, study participants should be supervised and any suspected adverse event (AE) will be addressed by the study dentist. There is a record of adverse events (Annex 11), where you can record any reaction such as: dental caries, premature contact points and allergy. In case of an adverse event (AE); the first contact will be with the dentist of the responsible study who is in the province of Pichanaki. Immediate tele-dentistry will be done to see the problem. It will be referred within 48 hours in the pertinent time. in dentistry, adverse problems are considered emergencies and not emergencies. The sponsor, school principal, parents, ethics committee, and study investigators will be informed.The progress of the clinical trial will be monitored every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children whose parents accepted their participation in the study and who signed the Informed Consent (Annex 1)
* Children enrolled in the school of the district of Pichanaki, province of Chanchamayo and department of Junín
* Children between 6 and 8 years, with permanent upper and / or lower molars with the following characteristics:

Deep cavities and cavities free of cavities, rated 0 and 1 according to ICDAS II Non-cavitated caries in enamel C1 according to ICDAS II Green and Vermillion Simplified Oral Hygiene Index (OHS) of 1 Have a pair of non-cavitated caries-free counterparts.

-Collaborative and receptive children.

Exclusion Criteria:

* Children with the presence of a deep dental caries lesion, with pulp exposure, history of pain and presence of fistula or abscess adjacent to decayed tooth.
* Medically compromised children
* Children with developmental enamel defects.
* Children with a known allergy to any of the resins used
* Children with previously placed sealants or restorations
* Children with bruxism or malocclusion
* Children residing outside the city.
* Children with poor hygiene

Criteria for withdrawal of research subjects

* When they did not attend the evaluations
* If the participant has partial retention and total loss of the sealant, he will be withdrawn from the study after placing a new sealant.
* If a patient moves to another region, it will be grounds for withdrawal from the study.
* If the patient wishes to leave the study, they are considered outside the study

Criteria for termination or interruption of the clinical trial.

* When the 12-month follow-up of all the recruited patients, excluding the withdrawn ones, is completed, the study will be terminated.
* Work is interrupted

Ages: 6 Years to 8 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Retention of sealants | 12 months
  Determine which of the two sealants has better retention during the period of 12 months, one based on flowable resin with sprg the other only based on flowable resin

SECONDARY OUTCOMES:
Clinical preservation | 12 months
  Evaluate of clinical preservation of a sealant based on flowable resin with sprg and another based on flowable resin in first permanent molars, in the period of 12 months
Survival curve | 12 months
  Estimate the survival curve of a sealant based on flowable resin with sprg and another based on flowable resin in first permanent molars, in the period of 12 months.
Survival of the sealant | 12 months
  Compare the survival of a sealant based on flowable resin with sprg and another based on flowable resin in first permanent molars, in the period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ruiz Yasuda, Doctor, Principal Investigator — Faculty of dentistry UNMSM.
Locations (1):
- Manuel Gonzales Prada School, Alto Pichanaki, Chanchamayo, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nayhua Gamarra L, Grados Soto F, Llallico Huancaya W, Portocarrero Pechiarovich J, Virhuez Díaz T, Cruz Martínez A, et al. Technical Document Epidemiological Profile of Oral Health in school children from 3 to 15 years old, Peru 2012-2014; 1-82
- [Background] Gillcrist JA, Vaughan MP, Plumlee GN Jr, Wade G. Clinical sealant retention following two different tooth-cleaning techniques. J Public Health Dent. 1998 Summer;58(3):254-6. doi: 10.1111/j.1752-7325.1998.tb03003.x. PMID 10101704
- [Result] de França TRT, Sedycias M, da Silva RJ, de Souza Beatrice LC, Vicente Da Silva CH. Use of Glass Ionomer Cement: A Systematic Review. Pesqui Bras Odontopediatria Clin Integr. 2010; 10 (2): 301-7.
- [Result] Provenzano, M. G. A., Rios, D., from Lourdes Calvo Fracasso, M., Marchesi, A., & Honório, H. M. Clinical Evaluation of Sealants Made with Resin Modified Glass Ionomer Cement (Vitremer®) in Primary Molars. Brazilian Research in Pediatric Dentistry and Integrated Clinic. 2010; 10 (2), 233-240.
- [Result] Hou J, Gu Y, Zhu L, Hu Y, Sun M, Xue H. Systemic review of the prevention of pit and fissure caries of permanent molars by resin sealants in children in China. J Investig Clin Dent. 2017 Feb;8(1). doi: 10.1111/jicd.12183. Epub 2015 Aug 14. PMID 26272130
- [Result] Topal BG, Kirzioglu Z. Evaluation of the fissure sealants applied to erupting permanent molars in accordance to eruption stages: A prospective study. Niger J Clin Pract. 2019 Nov;22(11):1495-1502. doi: 10.4103/njcp.njcp_534_18. PMID 31719270
- [Result] Minsa. Clinical practice guide for the prevention, diagnosis and treatment of dental caries in boys and girls.Resolution Minist N ° 422-2017 / MINSA [Internet]. 2017; 41.
- [Result] Alirezaei M, Bagherian A, Sarraf Shirazi A. Glass ionomer cements as fissure sealing materials: yes or no?: A systematic review and meta-analysis. J Am Dent Assoc. 2018 Jul;149(7):640-649.e9. doi: 10.1016/j.adaj.2018.02.001. Epub 2018 May 4. PMID 29735163
- [Result] Bagherian A, Shirazi AS. Flowable composite as fissure sealing material? A systematic review and meta-analysis. Br Dent J. 2018 Jan 26;224(2):92-97. doi: 10.1038/sj.bdj.2018.40. PMID 29372708
- [Result] Ministry of Health. National Center for Epidemiology, Disease Prevention and Control. Burden of disease in Peru: Estimation of healthy years of life lost 2016 part I. 2018; part I. Available from: https://www.gob.pe/institucion/minsa/informes-publicaciones/276778-carga-de -sickness-in-peru-estimate-of-healthy-years-of-life-lost-2016
- [Result] Ministry of Health: National Center for Epidemiology, Prevention and Control of Diseases. Estimation of healthy years of life lost 2016. Enferm Burden in Peru [Internet].2018; Part II: 22-44.
- [Result] Shimazu K, Ogata K, Karibe H. Evaluation of the ion-releasing and recharging abilities of a resin-based fissure sealant containing S-PRG filler. Dent Mater J. 2011;30(6):923-7. doi: 10.4012/dmj.2011-124. Epub 2011 Nov 25. PMID 22123018
- [Result] Abdel-karim UM, El-Eraky M, Etman WM. Three-year clinical evaluation of two nano-hybrid giomer restorative composites. Tanta Dent J [Internet]. 2014; 11 (3): 213-22.
- [Result] Kucukyilmaz E, Savas S. Evaluation of Different Fissure Sealant Materials and Flowable Composites Used as Pit-and-fissure Sealants: A 24-Month Clinical Trial. Pediatr Dent. 2015 Sep-Oct;37(5):468-73. PMID 26531092
- [Result] Ntaoutidou S, Arhakis A, Tolidis K, Kotsanos N. Clinical evaluation of a surface pre-reacted glass (S-PRG) filler-containing dental sealant placed with a self-etching primer/adhesive. Eur Arch Paediatr Dent. 2018 Dec;19(6):431-437. doi: 10.1007/s40368-018-0379-z. Epub 2018 Oct 16. PMID 30328064
- [Result] Wadhwa S, A Nayak U, Kappadi D, Prajapati D, Sharma R, Pawar A. Comparative Clinical Evaluation of Resin-based Pit and Fissure Sealant and Self-adhering Flowable Composite: An In Vivo Study. Int J Clin Pediatr Dent. 2018 Sep-Oct;11(5):430-434. doi: 10.5005/jp-journals-10005-1552. Epub 2018 Oct 1. PMID 30787558
- [Result] Yazici AR, Bayazit EO, Kutuk ZB, Ozgunaltay G, Ergin E, Berber A. Clinical Follow-up of a Fissure Sealant Placed Using Different Adhesive Protocols: A 24-month Split-mouth Study. Oper Dent. 2018 Jul/Aug;43(4):362-371. doi: 10.2341/17-055-C. Epub 2018 Apr 9. PMID 29630489
- [Result] Rishika, Garg N, Mayall SS, Pathivada L, Yeluri R. Combined Effect of Enamel Deproteinization and Intermediate Bonding in the Retention of Pit and Fissure Sealants in Children: A Randomized Clinical Trial. J Clin Pediatr Dent. 2018;42(6):427-433. doi: 10.17796/1053-4625-42.6.4. Epub 2018 Aug 7. PMID 30085876
- [Result] Papageorgiou SN, Dimitraki D, Kotsanos N, Bekes K, van Waes H. Performance of pit and fissure sealants according to tooth characteristics: A systematic review and meta-analysis. J Dent. 2017 Nov;66:8-17. doi: 10.1016/j.jdent.2017.08.004. Epub 2017 Aug 8. PMID 28797916
- [Result] Erdemir U, Sancakli HS, Yaman BC, Ozel S, Yucel T, Yildiz E. Clinical comparison of a flowable composite and fissure sealant: a 24-month split-mouth, randomized, and controlled study. J Dent. 2014 Feb;42(2):149-57. doi: 10.1016/j.jdent.2013.11.015. Epub 2013 Dec 1. PMID 24296163
- [Result] Jafarzadeh M, Malekafzali B, Tadayon N, Fallahi S. Retention of a Flowable Composite Resin in Comparison to a Conventional Resin-Based Sealant: One-year Follow-up. J Dent (Tehran). 2010 Winter;7(1):1-5. Epub 2010 Mar 31. PMID 21998768
- [Result] Cogo E, Calura G. Clinical evaluation of two materials Ußed As P I T and Fissure Sealants :2-year follow-up. International Journal of Clinical Dentistry Volume 2, Issue 4
- [Result] Khanna R, Pandey RK, Singh N . Morphology of Pits and Fissures Reviewed through Scanning Electron Microscope. Dentistry. 2015,5: 4. doi:10.4172/2161-1122.1000287
- [Result] Kimura M, Maki K, Nishida I, Braham RL. Clinical evaluation of a light-cured glass ionomer lining cement. Int J Paediatr Dent. 1994 Sep;4(3):147-50. doi: 10.1111/j.1365-263x.1994.tb00123.x. PMID 7811668
- [Result] Vaillard-Jiménez, E & Huitzil-Muñoz, E & Ortega, Ai & García-Damián S. Dimensional Characteristics of Fissures and Enamel Fissures of Temporary Molars. Rev Colomb Investig en Odontol [Internet]. 2013; 12 (2): 102-109. .
- [Result] Rechmann P, Charland D, Rechmann BM, Featherstone JD. Performance of laser fluorescence devices and visual examination for the detection of occlusal caries in permanent molars. J Biomed Opt. 2012 Mar;17(3):036006. doi: 10.1117/1.JBO.17.3.036006. PMID 22502564
- [Result] Diniz MB, Rodrigues JA, Hug I, Cordeiro Rde C, Lussi A. Reproducibility and accuracy of the ICDAS-II for occlusal caries detection. Community Dent Oral Epidemiol. 2009 Oct;37(5):399-404. doi: 10.1111/j.1600-0528.2009.00487.x. Epub 2009 Jul 22. PMID 19681984
- [Result] Van Meerbeek B, Yoshihara K, Van Landuyt K, Yoshida Y, Peumans M. From Buonocore's Pioneering Acid-Etch Technique to Self-Adhering Restoratives. A Status Perspective of Rapidly Advancing Dental Adhesive Technology. J Adhes Dent. 2020;22(1):7-34. doi: 10.3290/j.jad.a43994. PMID 32030373
- [Result] Muller-Bolla M, Lupi-Pegurier L, Tardieu C, Velly AM, Antomarchi C. Retention of resin-based pit and fissure sealants: A systematic review. Community Dent Oral Epidemiol. 2006 Oct;34(5):321-36. doi: 10.1111/j.1600-0528.2006.00319.x. PMID 16948671
- [Result] Espinosa R, Valencia R, Uribe M, Ceja I, Saadia M. Enamel deproteinization and its effect on acid etching: an in vitro study. J Clin Pediatr Dent. 2008 Fall;33(1):13-9. doi: 10.17796/jcpd.33.1.ng5462w5746j766p. PMID 19093646
- [Result] Duggal MS, Tahmassebi JF, Toumba KJ, Mavromati C. The effect of different etching times on the retention of fissure sealants in second primary and first permanent molars. Int J Paediatr Dent. 1997 Jun;7(2):81-6. doi: 10.1111/j.1365-263x.1997.tb00283.x. PMID 9524458
- [Result] Cobos-Carbo A, Augustovski F. [CONSORT 2010 Declaration: updated guideline for reporting parallel group randomised trials]. Med Clin (Barc). 2011 Jul 23;137(5):213-5. doi: 10.1016/j.medcli.2010.09.034. Epub 2011 Jan 15. No abstract available. Spanish. PMID 21239025
- [Result] National Institute of Health. (2017). Regulations for Clinical Trials are approved. El Peruano, pp. 38-67. Retrieved from https://ensayosclinicos-repec.ins.gob.pe/images/REC-021-2017-sa-1538902-2.pdf
- [Result] World medical association. Wma declaration of helsinki - ethical principles for medical investigations in human beings. 2017
- [Result] Pozos-Guillen A, Chavarria-Bolanos D, Garrocho-Rangel A. Split-mouth design in Paediatric Dentistry clinical trials. Eur J Paediatr Dent. 2017 Mar;18(1):61-65. doi: 10.23804/ejpd.2017.18.01.13. PMID 28494606
- [Result] Latin American Association of Pediatric Dentistry. Care Route for Pediatric Dental Procedures During the Confinement or Quarantine of the COVID-19 Pandemic: Dental EMERGENCY-URGENCY Consultation.2020; 10: 2-4.
- [Result] Mallineni SK, Innes NP, Raggio DP, Araujo MP, Robertson MD, Jayaraman J. Coronavirus disease (COVID-19): Characteristics in children and considerations for dentists providing their care. Int J Paediatr Dent. 2020 May;30(3):245-250. doi: 10.1111/ipd.12653. Epub 2020 Apr 16. PMID 32250505
- [Result] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Result] National cancer institute. NHI INFORMED CONSENT [Internet]. 2020 p. 163-6.
- [Result] Fejerskov O. Changing paradigms in concepts on dental caries: consequences for oral health care. Caries Res. 2004 May-Jun;38(3):182-91. doi: 10.1159/000077753. PMID 15153687
- [Result] Martignon S, Pitts NB, Goffin G, Mazevet M, Douglas GVA, Newton JT, Twetman S, Deery C, Domejean S, Jablonski-Momeni A, Banerjee A, Kolker J, Ricketts D, Santamaria RM. CariesCare practice guide: consensus on evidence into practice. Br Dent J. 2019 Sep;227(5):353-362. doi: 10.1038/s41415-019-0678-8. PMID 31520031
- See also: Use of Glass Ionomer Cement: A Systematic Review. Pesqui Bras Odontopediatria Clin Integr. 2010; 10 (2): 301-7. — https://www.redalyc.org/pdf/637/63716962025.pdf
- See also: Clinical Evaluation of Sealants Made with Resin Modified Glass Ionomer Cement (Vitremer®) in Primary Molars. Brazilian Research in Pediatric Dentistry and Integrated Clinic. 2010; 10 (2), 233-240. — https://pesquisa.bvsalud.org/gim/resource/en/lil-568484
- See also: Minsa. Clinical practice guide for the prevention, diagnosis and treatment of dental caries in boys and girls.Resolution Minist N ° 422-2017 / MINSA [Internet]. 2017; 41 — http://bvs.minsa.gob.pe/local/MINSA/4195.pdf
- See also: National Center for Epidemiology, Disease Prevention and Control. Burden of disease in Peru: Estimation of healthy years of life lost 2016 part I. 2018; part I. — https://cdn.www.gob.pe/uploads/document/file/315254/1.pdf
- See also: National Center for Epidemiology, Prevention and Control of Diseases. Estimation of healthy years of life lost 2016. Enferm Burden in Peru [Internet].2018; Part II: 22-44. — https://cdn.www.gob.pe/uploads/document/file/315255/2.pdf
- See also: Cogo E, Calura G. Clinical evaluation of two materials Ußed As P I T and Fissure Sealants :2-year follow-up. International Journal of Clinical Dentistry Volume 2, Issue 4 — http://www.novapublishers.org/catalog/product_info.php?products_id=19024
- See also: Regulations for Clinical Trials are approved. El Peruano, pp. 38-67. — https://ensayosclinicos-repec.ins.gob.pe/regulacion/normatividad-vigente/205-reglamento-de-ensayos-clinicos
- See also: World medical association. Wma declaration of helsinki - ethical principles for medical investigations in human beings. 2017 — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- See also: Vaillard-Jiménez, E & Huitzil-Muñoz, E & Ortega, Ai & García-Damián S. Dimensional Characteristics of Fissures and Enamel Fissures of Temporary Molars. Rev Colomb Investig en Odontol [Internet]. 2013; 12 (2): 102-109. — https://www.researchgate.net/publication/263419756_Caracteristicas_de_las_otras_formas_de_Nagano_de_fosas_y_fisuras_de_molares_temporales_Odontol_Pediatr_2013_122_102-109
- See also: Latin American Association of Pediatric Dentistry. Care Route for Pediatric Dental Procedures During the Confinement or Quarantine of the COVID-19 Pandemic: Dental EMERGENCY-URGENCY Consultation.2020; 10: 2-4 — https://odontologos.com.co/noticia/ruta-de-atencin-para-procedimientos-de-odontologa-peditrica-durante-la-etapa-de-confinamiento-o-cuarentena-de-la-pandemia-covid-19
- See also: National cancer institute. NHI INFORMED CONSENT [Internet]. 2020 p. 163-6 — https://www.cancer.gov/about-cancer/treatment/clinical-trials/patient-safety/informed-consent